CLINICAL TRIAL: NCT04263532
Title: Randomized Controlled Cross-Over Pilot Study of the Effectiveness of the Vector NIV Device in Hypercapnic COPD Patients With Expiratory Flow Limitation
Brief Title: Vector Efficacy Cross-Over Pilot Study
Status: Terminated | Type: Interventional
Why Stopped: Study discontinued due to shifted business priorities.
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SRC-HRC-VectorEFF-2018-10377
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Patients who meet inclusion criteria will be randomized in a 1:1 ratio to receive either standard non-invasive ventilation (NIV) (control) or Vector (Active) for the first 4 to 6-week treatment period, followed by the other treatment during the second 4 to 6 weeks (see figure 1). There will be two different patient cohort groups, patients that are current users of NIV and patients that are Naïve to NIV.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (4):
- Vector Device (NIV Current Users) (Experimental): Participants will use the Vector device with settings from the 3-hour Vector titration.
  Interventions: Device: Modified BiPAP A40 with Vector Algorithm (Vector)
- Standard of Care NIV (NIV Current Users) (Active Comparator): Participants will use a Vector Device in place of their current NIV device. The Vector therapy will not be enabled, and the device will be set according to their current standard of care NIV prescription.
  Interventions: Device: Modified BiPAP A40 with Standard of Care Settings
- Vector Device (NIV Naive) (Experimental): Participants will use the Vector device with settings from the 3-hour Vector titration.
  Interventions: Device: Modified BiPAP A40 with Vector Algorithm (Vector)
- Standard of Care NIV (NIV Naive) (Active Comparator): Participants will use the Vector device (Vector therapy will be enabled) with settings from a standard of care NIV titration.
  Interventions: Device: Modified BiPAP A40 with Standard of Care Settings

INTERVENTIONS:
Device: Modified BiPAP A40 with Vector Algorithm (Vector) — The Modified BiPAP A40 with Vector Algorithm (Vector) is intended to provide non-invasive ventilatory support to treat patients weighing over 10 kg (22 lbs) with Obstructive Sleep Apnea (OSA) or Respiratory Insufficiency. It is intended to be used within the home, institutional/ hospital, and diagnostic laboratory environments. This device is not intended for life support. The BiPAP A40 EFL screening and therapy is intended for patients weighing over 30 kg (66 lbs) with Obstructive Sleep Apnea (OSA), or Respiratory Insufficiency with primary cause being Chronic Obstructive Pulmonary Disease (COPD) to screen for the presence, and abolishment of Expiratory Flow Limitation (EFL).
  Arms: Vector Device (NIV Current Users); Vector Device (NIV Naive)
Device: Modified BiPAP A40 with Standard of Care Settings — The Modified BiPAP A40 with Standard of Care settings is intended to provide non-invasive ventilatory support to treat patients weighing over 10 kg (22 lbs) with Obstructive Sleep Apnea (OSA) or Respiratory Insufficiency. It is intended to be used within the home, institutional/ hospital, and diagnostic laboratory environments. This device is not intended for life support. The BiPAP A40 EFL screening and therapy is intended for patients weighing over 30 kg (66 lbs) with Obstructive Sleep Apnea (OSA), or Respiratory Insufficiency with primary cause being Chronic Obstructive Pulmonary Disease (COPD) to screen for the presence, and abolishment of Expiratory Flow Limitation (EFL).
  Arms: Standard of Care NIV (NIV Current Users); Standard of Care NIV (NIV Naive)

SUMMARY:
The study evaluates the safety and efficacy of the modified Bi-level positive airway pressure (BiPAP) A40 with Vector Algorithm to treat Chronic Obstructive Pulmonary Disease (COPD) patients with excessive carbon dioxide in their bloodstream (hypercapnia) and expiratory flow limitation (EFL), a constriction of the lower airways. The study will include current users of non-invasive ventilation (NIV) as well as those who are not currently using an NIV device.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled cross-over pilot trial to investigate the clinical efficacy and safety of the Modified Bi-level positive airway pressure (BiPAP) A40 with Vector Algorithm (Vector Device), a non-invasive ventilation (NIV) device, to treat Chronic Obstructive Pulmonary Disease (COPD). Approximately 30 COPD patients with chronic hypercapnia and evidence of expiratory flow limitation (EFL) will be included. It is estimated that 50 patients may need to be enrolled in order to complete 30. There will be two different patient cohort groups, patients that are current users of NIV and patients that are Naïve to NIV. Only those that meet the inclusion/exclusion criteria will be screened to determine if EFL is present. If participants are found to have EFL they will undergo a 20 minute EFL abolishment determination. Those participants that have EFL and a titrated expiratory positive airway pressure (EPAP) ≥6cmH2O will be scheduled for study visit 2. During study visit 2, participants will be randomized in a 1:1 ratio to receive either standard NIV (control) or Vector (Active) for the first 4 to 6-week at-home treatment period, followed by the other treatment during the second 4 to 6 weeks. Participants will have up to 4 (NIV current Users) or 5 (NIV Naïve) in-person visits that will include 2 overnight sleep studies with polysomnogram (PSG).

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 40 years of age; less than or equal to 80 years of age
2. Ability to provide consent
3. Chronic obstructive pulmonary disease (COPD) patients with hypercapnia (as defined as greater than or equal to 52mmHg) who are either current non-invasive ventilation (NIV) users or naïve to NIV
4. On average, use NIV more than 4 hours per night (Current NIV users).
5. Must present with expiratory flow limitation (EFL) via screening of the Vector device at 3 cmH2O
6. Have an EPAP to abolish EFL greater or equal to 6cmH2O

Exclusion Criteria:

1. Any major non-COPD uncontrolled disease or condition, such as congestive heart failure, malignancy, liver or renal insufficiency (that requires current evaluation for liver or renal transplantation or dialysis), amyotrophic lateral sclerosis, or severe stroke, or other condition as deemed appropriate by investigator as determined by review of medical history and / or participant reported medical history
2. Suffering from a COPD exacerbation (Defined as hospital admission, ER/urgent care visit, MD visit with medication change or other intervention deemed to be clinically significant by the investigator at the time of data collection or in the 14 days prior to data collection
3. Self-reported Pregnancy or positive pregnancy test for women of childbearing potential.
4. Employee or family member that is affiliated with Philips
5. Currently employed by a manufacturer of respiratory products or family member employed by a manufacturer of respiratory products
6. Any history of giant bulla (size >1/3 hemi-thorax)
7. History of pneumothorax < 6 months
8. Participants currently using a PAP or NIV device at home with a documented EPAP setting on their current device that is greater than the calculated EPAP determined during the therapy session of the screening visit (Current NIV Users).
9. Life expectancy ≤12 months as determined by clinical investigator
10. Low BP: Systolic <90
11. Recent cranial surgery (i.e, less than 1 year)
12. Impaired swallowing as reported by participant or diagnostic exam
13. Recent upper airway or GI surgery within the past 6 months
14. Unable to be fitted with mask
15. Excessive secretions as reported by clinical investigator/physician assessment, inability to maintain a patent airway or adequately clear secretions, or at risk for aspiration of gastric contents
16. Diagnosed with acute sinusitis or otitis media
17. Epistaxis, causing pulmonary aspiration of blood
18. Existing respiratory failure
19. Participants who are naïve to NIV (Cohort 2) that use the device fewer than 3 out of 7 nights during the second week of the 2-week acclimation period
20. Participants who are naïve to NIV (Cohort 2) that average less than 4 hours of device use during the second week of the 2-week acclimation period
21. Participants who are naïve to NIV (Cohort 2) with an average nightly 90% EPAP pressure during the second week of the 2-week acclimation period that is higher than the titrated EFL EPAP pressure determined at the screening visit.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 participants were consented and screened. 12 participants were screen failures, one of these participants was rescreened and determined to be eligible resulting in 10 participants being enrolled and randomized.
Groups:
- NIV Current Users: Vector, Then Standard of Care NIV: Experienced NIV participants assigned to the BiPAP A40 EFL device (Vector) for the first 4-6 week take home period followed by Standard of care for the second 4-6 week take home period.
- NIV Current Users: Standard of Care NIV, Then Vector: Experienced NIV participants assigned to the Standard of Care for the first 4-6 week take home period followed by BiPAP A40 EFL device (Vector) for the second 4-6 week take home period.
Period: Overall Study
Arm/Group | NIV Current Users: Vector, Then Standard of Care NIV | NIV Current Users: Standard of Care NIV, Then Vector
Started | 5 | 5
Completed | 3 | 5
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: 21 participants were consented and screened. 12 participants were screen failures, one of these participants was rescreened and determined to be eligible resulting in 10 participants being enrolled.
Groups:
- Randomized Participants: All participants that were enrolled and randomized.
- Screen Fails: All participants that were screen failed.
- Total: Total of all reporting groups
Arm/Group | Randomized Participants | Screen Fails | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (8.4) | 70.1 (4.7) | 66.7 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Daytime PaCO2 (Arterial Blood Gas)
Description: Room air CO2 levels at the end of 4-6 weeks of therapy as determined by Arterial Blood Gas (PaCO2)
Time Frame: At the end of the 4-to-6-week period
Population: 10 participants were randomized, 2 participants received Standard of care for both arms, so they were excluded from analysis, 2 additional participants discontinued prior to completing both arms and they were excluded from the analysis. 1 participant did not contribute PaCO2 data. No NIV naive participants were enrolled.
Measure: Mean (Standard Deviation); unit: mmHG
Groups:
- Vector Device (NIV Current Users): Experienced NIV participants assigned to the BiPAP A40 EFL device (Vector) for the 4-6 week take home period.
- Standard of Care NIV (NIV Current Users): Experienced NIV participants assigned to their Standard of care NIV prescription for the 4-6 week take home period. Participants will use a Vector Device in place of their current NIV device. The Vector therapy will not be enabled, and the device will be set according to their current standard of care NIV prescription.
Arm/Group | Vector Device (NIV Current Users) | Standard of Care NIV (NIV Current Users)
Number analyzed (Participants) | 5 | 5
mmHG | 59.2 (16.6) | 49.8 (8.8)

2. Secondary Outcome: Average 30 Day Ventilator Usage Hours
Description: How many hours per night over 30 days that the participant uses the device.
Time Frame: Up to 30 days of device use
Population: Processed data was only available N=3 participants. Average adherence was calculated among all days in the time period.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vector Device (NIV Current Users) | Standard of Care NIV (NIV Current Users)
Number analyzed (Participants) | 3 | 3
hours | 7.58 (4.52) | 7.40 (3.38)

3. Secondary Outcome: Patient Comfort and Therapy Preference Based Questionnaire Responses
Description: Comfort data from device satisfaction/preference questionnaire after 30 days of device use. The specific question analyzed was " Which ventilator pressure settings or therapy did you prefer?" Outcome was number of participants who selected each therapy as preferred.
Time Frame: Up to 30 days of device use
Population: 10 participants were randomized, 2 participants received Standard of care for both arms, and they were excluded from analysis, 2 additional participants discontinued prior to completing both arms and they were excluded from the analysis. The 6 participants answered comparative survey after completing both arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Vector Device (NIV Current Users) | Standard of Care NIV (NIV Current Users)
Number analyzed (Participants) | 6 | 6
Participants | 3 | 3

4. Secondary Outcome: Unanticipated Serious Adverse Device Effects (USADEs) and Serious Adverse Events (SAEs) Assessment
Description: Incidence of Unanticipated Serious Adverse Device Effects (USADEs) and Serious Adverse Events (SAEs) for the Vector vs. the control group.
Time Frame: Up to 30 days of device use
Population: Frequency of USADEs or SAEs when participant was using the assigned treatment. All SAEs which occurred were determined to be unrelated to the device. The term "incidence" in the protocol endpoint was imprecise. Frequency is the more appropriate term.
Measure: Count of Participants; unit: Participants
Arm/Group | Vector Device (NIV Current Users) | Standard of Care NIV (NIV Current Users)
Number analyzed (Participants) | 10 | 10
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: Approximately 15 weeks.
Groups:
- NIV Current Users: Vector: Experienced NIV participants assigned to the BiPAP A40 EFL device (Vector) for a 4-6 week take home period.
- NIV Current Users: Standard of Care NIV: Experienced NIV participants assigned to the Standard of Care for a 4-6 week take home period.
Arm/Group | NIV Current Users: Vector | NIV Current Users: Standard of Care NIV
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NIV Current Users: Vector (N=10) | NIV Current Users: Standard of Care NIV (N=10)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shortness of Breath and left sided chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypervolemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Presented with dyspnea on exertion, orthopnea, and bendopnea
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NIV Current Users: Vector (N=10) | NIV Current Users: Standard of Care NIV (N=10)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abnormal Blood gas level (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT04263532/Prot_SAP_000.pdf